CLINICAL TRIAL: NCT05411341
Title: Assessment of Two Different Optical Biometric Systems, Based on Different Optical Technologies in Patients With Cataract or Presbyopia
Brief Title: Comparison of Two Different Optical Biometric Systems
Status: Recruiting | Type: Observational
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Professor (Associate) of Democritus University of Thrace, Democritus University of Thrace
Other Study IDs: ES9/Th3/05-05-2022
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Cataract; Presbyopia; Ocular Biometry; Intraocular Lens
Keywords: cataract; presbyopia; argos; iol master 500; optical biometric system
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: 100 patients with diagnosed cataract or presbyopia who will undergo implantation of intraocular lenses surgery
  Interventions: Device: Argos (Alcon Laboratories, Inc.); Device: IOLMaster 500 (Carl Zeiss Meditec AG)

INTERVENTIONS:
Device: Argos (Alcon Laboratories, Inc.) — An ocular biometry examination will be performed on the affected eyes using the Argos device.
Device: IOLMaster 500 (Carl Zeiss Meditec AG) — An ocular biometry examination will be performed on the affected eyes using the IOL Master 500 device.

SUMMARY:
Primary objective of this study is to evaluate and compare the measurements of two different optical biometrics systems in patients who will undergo cataract surgery or presbyopia surgery using intraocular lenses (IOL-PC).

DETAILED DESCRIPTION:
This is a prospective study including patients visiting the outpatient Ophthalmology clinic of the University General Hospital of Alexandroupolis, who suffer from diagnosed cataract or presbyopia and are going to undergo implantation of intraocular lenses surgery. The patients will be fully informed about the procedure and the purpose of the study and a written informed consent will be provided by all participants. They will then undergo an ocular biometry examination using two optical biometric systems, Argos (Alcon Laboratories, Inc.) and IOLMaster 500 (Carl Zeiss Meditec AG). IOL Master 500 (Carl Zeiss Meditec AG) is a non-invasive optical biometer that uses partial coherence interferometry (PCI) with a wavelength of 780 nm to measure the AL of the eye. Argos (Alcon Laboratories, Inc.) is a novel non-invasive optical biometer that uses swept source optical coherence tomography (SS-OCT) with a wavelength of 1050 nm. The measurements of the two systems that will be compared are the axial length, the keratometry values, the anterior chamber depth (ACD), the horizontal corneal diameter (white to white [WTW]) and the lens power in diopters (D).

ELIGIBILITY:
Inclusion Criteria:

* Patients with cataract and/or presbyopia who will undergo intraocular lens implantation.

Exclusion Criteria:

* Dense cataract that does not allow measurements to be taken with an optical biometrics system.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with cataract and/or presbyopia.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Axial length | 1 week
  The measurement of the axial length of the affected eye using both devices
Keratometry values | 1 week
  The measurement of keratometry values K1: flat meridian of the anterior corneal surface and K2: steep meridian of the anterior corneal surface of the affected eye using both devices.
Lens power (D) | 1 week
  The power of the lens is calculated by each device as a function of biometric measurements

SECONDARY OUTCOMES:
Anterior chamber depth (ACD) | 1 week
  The measurement of the anterior chamber depth (ACD) of the affected eye using both devices.
Horizontal corneal diameter (white to white [WTW]) | 1 week
  The measurement of the horizontal corneal diameter of the affected eye using both devices.

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, MD, PhD, Study Chair — Department of Ophthalmology, University Hospital of Alexandroupolis, Alexandroupolis, Greece
Locations (1):
- Department of Ophthalmology, University Hospital of Alexandroupolis, Alexandroupoli, Evros, Greece